CLINICAL TRIAL: NCT02014233
Title: The Effect of Short Term Omega-3 Supplementation on Exercise Performance and Neuromuscular Function.
Brief Title: Short Term Omega-3 Supplementation on Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Thomas Wolever, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: UTTW-N3-1
Record Dates: First submitted 2013-10-25; First posted 2013-12-18 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Muscle Fatigue; Muscle Strength
Keywords: Randomized clinical trial; Humans; Omega-3 fatty acids; Essential fatty acid; Neuromuscular function; Wingate; Maximum voluntary contraction; Electromyography; Seal oil; Cycling time trial; Placebo controlled
MeSH Terms: interventions — Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 (Experimental): Participants will consume 5 mL of omega-3 (2333 mg essential fatty acids) with 1000 IU vitamin D3 for 21 days.
  Interventions: Dietary Supplement: Omega-3
- Olive oil (Placebo Comparator): Participants will consume 5 mL of olive oil with 1000 IU vitamin D3 for 21 days.
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Omega-3
  Other Names: Auum Omega Sublingual D; NPN 80014581
  Arms: Omega-3
Dietary Supplement: Olive oil
  Arms: Olive oil

SUMMARY:
Nerves are the rate limiting factor that control muscle function. However, it is unknown if a nutritional supplement can change the nerve-muscle interaction, and therefore alter human performance. This study will be the first to examine the effects of omega-3 supplementation on neuromuscular function in trained individuals.

DETAILED DESCRIPTION:
Participants will come to the lab for 3 sessions, one for familiarization and two for testing.

Familiarization - At this time, anthropometric measurements including height, weight, BMI (body mass index) and body composition will be determined. Participants will be familiarized with the interpolated twitch technique and performing a maximal voluntary contraction of the quadriceps muscle. Next, Participant's 10 repetition maximum squat weight will be established by starting at a participant selected weight and gradually increasing until only 10 squat repetitions can be completed. A VO2max (maximum oxygen consumption) test will be performed on a cycle ergometer using standard methods.

On testing sessions 1 and 2 the following neuromuscular and performance measures will be evaluated:

1. Quadriceps muscle voluntary activation will be assessed using the interpolated twitch technique and doublet twitch technique. Participants will be seated and instructed to perform three 5 second maximal voluntary isometric contractions at least 1 minute apart - participant's ankle will be restrained by a padded cuff attached to a load cell.

   For the second maximal isometric contraction at 3 seconds into the contraction, a square wave superimposed stimulus will be delivered for 1 milliseconds to the femoral nerve from a monopolar touch-proof cathode electrode secured in the femoral triangle. 2, 7 and 12 seconds after the contraction a resting twitch will be delivered for comparison of muscle force.

   For the third maximal isometric contraction, at 3 seconds into the contraction, two 1 millisecond square wave superimposed stimuli at 100 Hz will be delivered 10 milliseconds apart. 2 seconds after the contraction the same stimulus will be applied. At 7 seconds after, two stimuli will be delivered 100 milliseconds at 10 Hz apart and 12 seconds after a single stimulus will be delivered.

   The percutaneous electrical stimulation will be delivered from a Biopac stimulator (BSLSTMA, Biopac Systems, Santa Barbara, California) with a maximum voltage of 400 V. During familiarization, participants will receive several submaximal stimulations for acclimatization before the current intensity is gradually increased until peak twitch torque and muscle action potential amplitude is reached. A stimulus of 1.2 times the current required to elicit peak twitch torque and action potential amplitude will be used to ensure maximal activation. The interpolated twitch technique will be used to examine the difference in muscle activation during maximal contraction and a superimposed stimulation. Voluntary activation will be calculated using the formula:

   Voluntary activation (%) = (1- superimposed twitch / twitch evoked at rest) x 100

   Surface self-adhesive silver chloride electrodes will be placed over the belly of the vastus lateralis, vastus medialis and biceps femoris muscles to measure muscle electrical activity (electromyography) during maximal voluntary contractions as previously described.
2. Vertical jump - Quadriceps power will be assessed using the vertical jump test on a force plate (AMTI, Watertown, Massachusetts, USA). Participants will complete two attempts to jump as high as possible from crouched and two attempts using the counter jump technique (participants can start from standing, bend the knees and then jump).
3. Push-up - Upper body strength endurance will be examined by having the participant complete as many push-ups as possible in one-minute. Participants will be given one-minute rest before being asked to complete as many push-ups as possible in a minute. A piece of soft foam will be attached to the floor to provide participants feedback as to how low the must go when performing each push-up.
4. 10RM (10 repetition maximum) squat - After completing an optional 2 to 4 repetitions of 75% of the their 10RM weight as determined during baseline data collection, participants will complete as many repetitions as possible.
5. Wingate test - Participants will be fitted to a cycle ergometer (Excalibur Sport V2.0, Lode, Groningen, The Netherlands). They will then cycle against a fixed resistance of 0.075kg / kg body mass for 30 seconds using their maximum effort. Verbal encouragement will be provided to the participant to help produce their maximum effort.
6. Cycling time trial - Participants will complete a 10km time trial on a cycle ergometer (Excalibur Sport V2.0, Lode, Groningen, The Netherlands). Participants' inspired and expired gasses will be measured using a metabolic cart (Cortex, Leipzig, Germany). Gas variables and cycling power output will be measured using the supplied software. This change in protocol does not alter the risk to participants as their level of conditioning is quite high and similar levels of exertion would be required in their daily training.

Supplementation - In between sessions 1 and 2, there is a 21 day break for which participants will be computer randomized to either the omega-3 supplementation or an olive oil placebo. Participants will take a 2.5 mL serving of seal oil (2500 mg n-3, 255 mg DHA (docosahexaenoic acid ) and 187.5 mg EPA (eicosapentaenoic acid) with 500 IU vitamin D3 and 1000 IU vitamin A) (Auum Inc., Timmons, On) or 2.5 mL olive oil (Bertolli, Mississauga, Ont) with 500 IU vitamin D and 1000 IU vitamin A added twice daily with breakfast and dinner.

All supplementation amounts are within the amounts specified by Health Canada Guidelines.

Session 2 - After the 21 day supplementation period, participants will return to the lab for a second evaluatory session using identical protocols to session 1.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 years training experience that includes resistance training, specifically back squat
* Successfully completing a Par-Q questionnaire

Exclusion Criteria:

* Individuals that have or are currently taking an omega-3 and/or omega-6 supplement within 4 weeks of the study
* Individuals that have taken mammalian based omega-3 or 6 supplements in the past 6 months
* Individuals consuming fish more than twice per week within 4 weeks of the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in maximum voluntary contraction force | 21 days
  Participants will be seated with their right knee fixed at 90°. The right ankle will be restrained by a padded cuff attached in series to a load cell. Participants will be instructed to contract their quadriceps maximally by trying to extending their leg. The load cell will measure the maximum force produced.

SECONDARY OUTCOMES:
Change from baseline in vertical jump height | 21 days
  Participants will perform both squat jumps and counter movement jumps on a force plate. Jump height (cm) will be measured.
Change from baseline in number of push-ups | 21 days
  Participants will perform the maximum number of push-ups possible in one minute while maintaining proper form. A one minute rest will be given and then they will repeat the same procedure.
Change from baseline in number of 10RM squats | 21 days
  Participants will complete as many reps of back squats possible using the 10 repetition maximum weight established during familiarization.
Change from baseline in Wingate test peak power | 21 days
  Participants will perform a 30 second maximal cycling sprint with the resistance set at 7.5% of their baseline body weight. Peak power, average power, fatigue index and cadence will all be measured.
Change from baseline in 250 kJ cycling time trial time to completion | Baseline and 21 days
  Participants will complete 250 kJ (kilo Joules) of cycling on an ergometer which is equivalent to 10km. Time to completion and average power (Watts) will be measured.
Change from baseline in Pre/Post maximal voluntary contraction force | 21 days
  Pre/Post quadriceps maximal voluntary contraction force is the difference in maximal voluntary contraction force measured at the beginning and end of each testing session to determine changes in neuromuscular function as a result of the other fatiguing tests.
Change from baseline in quadriceps voluntary activation | 21 days
  Participants femoral nerve will be electrically stimulated during the maximal voluntary contraction. Voluntary activation is the difference in muscle force output between the voluntary contraction and the electrically stimulated contraction.
Change from baseline in Wingate test average power | 21 days
  Participants will perform a 30 second maximal cycling sprint with the resistance set at 7.5% of their baseline body weight. Peak power, average power, fatigue index and cadence will all be measured.
Change from baseline in Wingate test fatigue index | 21 days
  Participants will perform a 30 second maximal cycling sprint with the resistance set at 7.5% of their baseline body weight. Peak power, average power, fatigue index and cadence will all be measured.
Change from baseline in Wingate test cadence | 21 days
  Participants will perform a 30 second maximal cycling sprint with the resistance set at 7.5% of their baseline body weight. Peak power, average power, fatigue index and cadence will all be measured.
Change from baseline in 250 kJ cycling time trial average power | Baseline and 21 days
  Participants will complete 250 kJ of cycling on an ergometer which is equivalent to 10km. Time to completion and average power (Watts) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Millet GY, Tomazin K, Verges S, Vincent C, Bonnefoy R, Boisson RC, Gergele L, Feasson L, Martin V. Neuromuscular consequences of an extreme mountain ultra-marathon. PLoS One. 2011 Feb 22;6(2):e17059. doi: 10.1371/journal.pone.0017059. PMID 21364944
- [Background] Presland JD, Dowson MN, Cairns SP. Changes of motor drive, cortical arousal and perceived exertion following prolonged cycling to exhaustion. Eur J Appl Physiol. 2005 Sep;95(1):42-51. doi: 10.1007/s00421-005-1395-3. Epub 2005 Jun 23. PMID 15976997
- [Background] Rodacki CL, Rodacki AL, Pereira G, Naliwaiko K, Coelho I, Pequito D, Fernandes LC. Fish-oil supplementation enhances the effects of strength training in elderly women. Am J Clin Nutr. 2012 Feb;95(2):428-36. doi: 10.3945/ajcn.111.021915. Epub 2012 Jan 4. PMID 22218156
- [Background] MERTON PA. Voluntary strength and fatigue. J Physiol. 1954 Mar 29;123(3):553-64. doi: 10.1113/jphysiol.1954.sp005070. No abstract available. PMID 13152698
- [Background] Behm DG, St-Pierre DM, Perez D. Muscle inactivation: assessment of interpolated twitch technique. J Appl Physiol (1985). 1996 Nov;81(5):2267-73. doi: 10.1152/jappl.1996.81.5.2267. PMID 8941554